CLINICAL TRIAL: NCT02981095
Title: Bupivacaine Application Reduces Postthyroidectomy Pain: Cerrahpaşa Experience
Brief Title: Effect of Bupivacaine Application on Postthyroidectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Serkan TEKSOZ, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUCTF-EndSx-2010-01
Record Dates: First submitted 2016-11-25; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Thyroid Disease; Analgesia
MeSH Terms: conditions — Thyroid Diseases; Agnosia | interventions — Thyroidectomy; Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): bupivacaine 0.5%, 10cc was administered to surgical field after completion of Thyroidectomy and approximately 15-30 minutes before the extubation.
  Interventions: Procedure: Thyroidectomy; Drug: Bupivacaine
- Saline (Placebo Comparator): Saline solution (%0.9 sodium chloride), 10cc was administered to surgical field after completion of Thyroidectomy and approximately 15-30 minutes before the extubation.
  Interventions: Procedure: Thyroidectomy; Drug: Saline Solution

INTERVENTIONS:
Procedure: Thyroidectomy — Thyroidectomy performed by the same surgical and anesthesia team
Drug: Bupivacaine — bupivacaine 0.5%, 10cc was administered to surgical field after completion of Thyroidectomy and approximately 15-30 minutes before the extubation.
  Arms: Bupivacaine
Drug: Saline Solution — %0.9 sodium chloride solution, 10cc was administered to surgical field after completion of Thyroidectomy and approximately 15-30 minutes before the extubation.
  Arms: Saline

SUMMARY:
Investigators aimed to evaluate the impact of bupivacaine administration into the surgical field after total thyroidectomy on post-operative pain and analgesic requirement with a double-blind, prospective, clinical, randomized study.

Pain assessment was performed with the visual analog score (VAS). Participants were pre-operatively, divided into two groups randomly to receive either bupivacaine or not. One group received a 10 ml of bupivacaine solution while the other group was treated with the same volume of 0.9% sodium chloride (NaCl) through the drain after completion of total thyroidectomy procedure. All participants were anesthetized and operated with the same anesthesia and surgical team.

ELIGIBILITY:
Inclusion Criteria:

* Subjects need to be operated for thyroid diseases

Exclusion Criteria:

* History of previous thyroid disease,
* History of previous neck operations,
* Hypersensitivity to the drugs that were used in the study protocol,
* Spinal bone disease,
* Depression,
* Kidney failure,
* Heart failure,
* Liver failure,
* Pulmonary failure,
* Mental retardation,
* Subjects not able to ascertain pain scoring with the visual analog score (VAS),
* Patients with American Society of Anesthesiologists (ASA) scores III or higher,
* Expected airway difficulty according to Mallampati scores,
* Sedative, steroid, and chronic analgesic drug users,
* Alcoholics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Post-operative pain in 8 hours after surgery using VAS | 8th hour
  Evaluation of the pain through the post-operative first 8 hours using VAS

SECONDARY OUTCOMES:
Post-operative pain in in first post-operative day using VAS | 1 day
  Evaluation of the pain through the first post-operative day using VAS

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf BUKEY, Prof. MD, Study Chair — Istanbul University
Locations (1):
- Istanbul University, Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No